CLINICAL TRIAL: NCT01238965
Title: Phase I Clinical Trial With LBH589 and Infusional 5-FU/LV in Patients With Metastatic Colorectal Cancer Who Failed 5-FU Based Chemotherapy
Brief Title: Panobinostat and Fluorouracil Followed By Leucovorin Calcium in Treating Patients With Stage IV Colorectal Cancer Who Did Not Respond to Previous Fluorouracil-Based Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adverse Events
Sponsor: University of Southern California (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-08-1; NCI-2010-02149
Record Dates: First submitted 2010-11-03; First posted 2010-11-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Panobinostat; Fluorouracil; Leucovorin; Biopsy; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral panobinostat 3 times a week. Patients also receive leucovorin calcium IV over 2 hours on days 1 and 15 followed by fluorouracil IV continuously over 46 hours on days 1-2 and 15-16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: panobinostat; Drug: fluorouracil; Drug: leucovorin calcium; Procedure: biopsy; Genetic: reverse transcriptase-polymerase chain reaction; Genetic: western blotting; Other: laboratory biomarker analysis; Genetic: gene expression analysis; Genetic: RNA analysis; Genetic: polymorphism analysis

INTERVENTIONS:
Drug: panobinostat — Given orally
  Other Names: Faridak; HDAC inhibitor LBH589; histone deacetylase inhibitor LBH589; LBH589
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU; Adrucil; Efudex; FU
Drug: leucovorin calcium — Given IV
  Other Names: calcium folinate; CF; CFR; citrovorum factor; LV; Wellcovorin
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Other: laboratory biomarker analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies
Genetic: RNA analysis — Correlative studies
Genetic: polymorphism analysis — Correlative studies

SUMMARY:
Panobinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving panobinostat together with fluorouracil and leucovorin calcium may kill more tumor cells. PURPOSE: This phase I trial is studying the side effects and the best dose of giving panobinostat, fluorouracil, and leucovorin calcium together in treating patients with stage IV colorectal cancer who did not respond to previous fluorouracil-based chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of combining LBH589 with infusional 5-FU chemotherapy in the treatment of Stage IV colorectal cancer patients who have progressed on standard 5-FU regimens.

II. To determine the efficacy of LBH589 alone to produce consistent decreases in tumor thymidylate synthase (TS) expression.

SECONDARY OBJECTIVES:

I. To determine the time to tumor progression, progression free and overall survival of patients with advanced or metastatic colorectal cancer treated with LBH589 combined with infusional 5-FU.

II. To determine if TS repression by LBH589 predicts response to the combination of LBH589 and infusional 5-FU in patients who have already progressed on standard regimens containing 5-FU.

III. To obtain preliminary data on gene expression levels of TS, DPD and TP as well as germline polymorphisms of TS being associated with clinical outcome and toxicity.

IV. To obtain preliminary data on acetylation on peripheral blood mononuclear cells to establish biological activity in these patients at time of biopsies.

OUTLINE: Patients receive oral panobinostat 3 times a week. Patients also receive leucovorin calcium IV over 2 hours on days 1 and 15 followed by fluorouracil IV continuously over 46 hours on days 1-2 and 15-16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced/metastatic colorectal cancer
* Must have measurable disease
* Must have received prior therapy (in any setting) with 5-FU, CPT-11, and oxaliplatin; (may have received prior erbitux and bevacizumab, but it is not required)
* Must have received at least one prior chemotherapy regimen for advanced disease
* Tumor must be accessible for core biopsy at the beginning of treatment and patients have a high intratumoral TS expression level prior to the beginning of treatment
* Life expectancy of > 12 weeks
* ECOG performance status 0-2 (Karnofsky >= 50%)
* Normal organ and marrow function as defined below:
* Serum albumin >= 3g/dL
* AST/SGOT and ALT/SGPT =< 2.5 x upper limit of normal(ULN)or =< 5.0 x ULN if the transaminase elevation is due to liver metastasis
* Serum bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN or 24-hr creatinine clearance >= 50 ml/min
* Serum potassium >= LLN
* Serum phosphorous >= LLN
* Serum total calcium (corrected for serum albumin) or serum ionized calcium >= LLN
* Serum magnesium >= LLN
* TSH and free T4 within normal limits(WNL)(patients may be on thyroid hormone replacement)
* Leukocytes >= 3,000/μL
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Hemoglobin >= 9 mg/dL
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of LBH589 will be determined following review by the Principal Investigator
* Ability to understand and willing to sign a written informed consent document
* INR is =< 1.5 times ULN unless receiving therapeutic anticoagulation
* Patient is highly unlikely to conceive as indicated by at least one "yes" answer to the following questions:

  1. patient is a male and agrees to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication;
  2. surgically sterilized female;
  3. postmenopausal female >= 45 years of age with > 2 years since last menses;
  4. non-sterilized premenopausal female and agrees to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study and for 30 days after the last dose of study medication
* Baseline MUGA must demonstrate LVEF >= the lower limit of the institutional normal
* Clinically euthyroid; Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism

Exclusion Criteria:

* Male patients whose sexual partners are WOCBP not using effective birth control
* May not have received any other investigational agents within 28 days of study entry (chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy).
* May not receive other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study
* Patients with known brain metastases are excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LBH589; including sodium butyrate, trichostatin A (TSA), trapoxin (TPX), MS-27-275 and depsipeptide
* Severe and/or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding or patients of reproductive potential not using two effective methods of birth control; women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589
* History of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
* Unresolved diarrhea > CTCAE grade 1
* Acute infection requiring intravenous antibiotic, antiviral, or antifungal medications within 2 weeks prior to the start of study drugs
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C
* Screening ECG with a QTc > 450 msec
* Patients with congenital long QT syndrome
* History of sustained ventricular tachycardia
* Any history of ventricular fibrillation or torsades de pointes
* Bradycardia defined as heart rate < 50 beats per minute; patients with a pacemaker and heart rate >= 50 beats per minute are eligible
* Myocardial infarction or unstable angina within 6 months of study entry
* Congestive heart failure (NY Heart Association class III or IV)
* Right bundle branch block and left anterior hemiblock (bifascicular block)
* Prior cancer treatment with an HDAC inhibitor (e.g., vorinostat, Depsipeptide, MS-275, LAQ-824, PXD-101, and valproic acid)
* Uncontrolled hypertension
* Concomitant use of drugs with a risk of causing torsades de pointes
* Any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
* Patients needing valproic acid for any medical condition during the study or within 5 days prior to first LBH589

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety of this regimen | Up to 12 months

SECONDARY OUTCOMES:
Time to progression | At 3, 6, 9, and 12 months
Overall response rate | Every 2 months until disease recurrence or progression
Overall survival | At 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States